CLINICAL TRIAL: NCT01307124
Title: A Multicenter Randomized Study to Compare the Safety and Efficacy of Low-dose Versus Standard Dose Lopinavir/Ritonavir Containing HAART Regimen in Virological Suppressed HIV-infected Thai Children
Brief Title: Pediatric Study for Appropriate Dose of Ritonavir Boosted Lopinavir in Thai HIV-infected Children (PEARL)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Chulalongkorn University (Other); Queen Sirikit National Institute of Child Health (Other Government); Srinagarind Hospital, Khon Kaen University (Other); Bamrasnaradura Infectious Diseases Institute (Other Government); Nakornping Hospital (Other); Prapokklao Hospital (Unknown); Surin Hospital (Unknown); Sappasitthiprasong Hospital (Unknown); UdonThani Hospital (Other Government); Buddhachinaraj Hospital (Other); Phrachomklao Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HIV-NAT 152
Record Dates: First submitted 2011-02-03; First posted 2011-03-02 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: HIV-infected Children
Keywords: safety and efficacy; low dose LPV/r; standard dose LPV/r; HIV infected children
MeSH Terms: interventions — lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard dose (Active Comparator): Arm 1:LPV/r Standard dose BW 25-35 kg 300/75 mg BW >35-50 kg 400/100 mg
  Interventions: Drug: kaletra
- low dose (Experimental): Arm 2:Low dose BW 25-35 kg 200/50 mg BW >35-50 kg 300/75 mg
  Interventions: Drug: kaletra

INTERVENTIONS:
Drug: kaletra — The study participants will receive Lopinavir/ritonavir heat-stable tablet (100/25 mg or 200/50 mg) q 12 hour plus NRTIs. The other NRTIs is depend on physician discretion.
  Arm 1:LPV/r Standard dose Arm 2:Low dose BW 25-35 kg 300/75 mg 200/50 mg BW >35-50 kg 400/100 mg 300/75 mg

SUMMARY:
To compare the safety and efficacy of low-dose versus standard dose lopinavir/ritonavir containing HAART regimen in virological suppress, HIV RNA viral load < 50 copies/ml at 48 week

ELIGIBILITY:
Inclusion Criteria:

1. HIV infection children age < 18 years old
2. Currently on PI regimens
3. HIV RNA viral load < 50 copies/ml at screening
4. BW 25-50 kg
5. Written informed consent

Exclusion Criteria:

1. Relevant history or current condition of PI resistance, plasma HIV RNA > 1000 copies/ml after received the PI regimens for at least 6 months
2. On rifampin, nevirapine, efavirenz which have drug interaction with lopinavir
3. On double boosted protease inhibitors

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 199 (Actual)
Dates: Start 2011-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
To compare the safety and efficacy of low-dose versus standard dose lopinavir/ritonavir containing HAART regimen in virological suppress, HIV RNA viral load < 50 copies/ml at 48 week | 48 week
  proportion of patient who had HIV RNA < 50 copies/ml Safety issue: patient who had HIV RNA > 50 copies/ml during the study period will be checked for LPV blood level, if the LPV Cmin < 1 ug/ml. The dose of LPV/r will be adjusted to appropriate dose.

CONTACTS AND LOCATIONS:
Overall Officials: Thanyawee Puthanakit, MD, Principal Investigator — Department of Pediatric , Faculty of Medicine, Chulalongkorn University and Thai Red Cross AIDS Research Centre - HIV-NAT
Locations (10):
- Thailand (10):
  - Srinagarind Hospital, Khon Kaen University, Khon Kaen, Changwat Khon Kaen
  - Bamrasnaradura Institute, Nonthaburi, Changwat Nonthaburi
  - Queen Sirikit National Institute of Child Health, Bangkok
  - Prapokklao Hospital, Chanthaburi
  - Nakornping Hospital, Chiang Mai
  - Phrachomklao Hospital, Phetchaburi
  - Buddhachinaraj Hospital, Phitsanulok
  - Surin Hospital, Surin
  - Sappasitthiprasong Hospital, Ubonratchathani
  - Udonthani Hospital, Udon Thani

REFERENCES:
- [Result] A randomized study comparing low dose versus standard dose lopinavir/ritonavir among HIV-infected children with virological suppression . Presented at 7th IAS 2013 in June 30-July 3, 2013 in Kuala Lumpur, Malaysia as abstract presentation.
- [Result] Association of SCLO1B1 polymorphism and plasma concentration of lopinavir in HIV-infected children. Presented at 7th IAS 2013 in June 30-July 3, 2013 in Kuala Lumpur, Malaysia as abstract presentation and 5th International Workshop on HIV Pediatrics in June 28-29, 2013 in Kuala Lumpur, Malaysia
- See also: HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org